CLINICAL TRIAL: NCT04755894
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of Fixed-dose Combination of HDDO-1756 or Loose Combination of HDDO-17561/HDDO-17562 in Healthy Adult Volunteers
Brief Title: HDDO-1756 Bio Equivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HT-013-01
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental)
  Interventions: Drug: HDDO-1756
- group B (Active Comparator)
  Interventions: Drug: HDDO-17561/HDDO-17562

INTERVENTIONS:
Drug: HDDO-1756 — single dose
  Arms: group A
Drug: HDDO-17561/HDDO-17562 — single dose
  Arms: group B

SUMMARY:
For healthy adult volunteers, safety and pharmacokinetic properties are compared between the two formulations in the case of HDDO-1756 alone administration and HDDO-17561/HDDO-17562 combined administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 or older during screening
2. A person who weighs more than 50.0 kg and has a BMI of 18.0 kg/m2 or less and 30.0 kg/m2 or less.

   ☞ BMI (kg/m2) = Weight (kg) / {Long (m)}2
3. A person who has no chronic disease or medical treatment and has no pathological symptoms or findings as a result of an internal examination;
4. A person who has been determined to be eligible for a clinical trial according to the characteristics of the drug during screening, such as serum tests, hematologic tests, hematological tests, urine tests, urine tests, etc. and vital signs (physical tests) and 12-lead ECG tests.

Exclusion Criteria:

1. Current or past history of clinically significant liver, kidney, nervous system, respiratory system, endocrine system, blood and tumor, urinary system, cardiovascular system, digestive system, musculoskeletal disease, or mental illness, as well as those with the following symptoms or history:
2. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
3. Persons with a history of gastrointestinal diseases (cron disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (except simple appendectomy or hernia surgery) that may affect the absorption of drugs;

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic evaluation variables | 0~96 hours
  Cmax
pharmacokinetic evaluation variables | 0~96 hours
  AUC

CONTACTS AND LOCATIONS:
Locations (1):
- Hyundai Pharm, Seoul, South Korea